CLINICAL TRIAL: NCT02340494
Title: An Online Enhanced Education Tool for Young Women Newly Diagnosed With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WomensCHCanada
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Education; Breast Neoplasms; Internet; Health Resources
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Women without access to the website.
- Intervention group (Experimental): Women with access to the website.
  Interventions: Behavioral: Online Enhanced Education Tool

INTERVENTIONS:
Behavioral: Online Enhanced Education Tool — The website resource will be credible, comprehensive, relevant and engaging information that young women with breast cancer will use intensively for self-management and education.
  Arms: Intervention group

SUMMARY:
This project proposes to develop and test an internet resource - a supported self-management website - that will guide younger women to relevant knowledge and resources, and provide tools that will help YWBC become more skilled and confident in coping with the many challenges of breast cancer. The study will be conducted in collaboration with the newly funded, pan-Canadian Young Breast Cancer Cohort (CYBCC) program being led from Women's College Hospital. The resource is expected to reduce knowledge gaps experienced by YWBC, and help them be partners in decision-making about their care, which has been shown to reduce anxiety and depression years later.

DETAILED DESCRIPTION:
Women age 40 years and younger account for 5.4% of new breast cancer diagnoses in Canada, but suffer more negative impacts than older women, due to having a worse prognosis, more intensive treatment and greater physical, social, and emotional sequelae due to life-stage factors. Consequently, younger women experience poorer quality of life, more problematic psychosocial adjustment to breast cancer and report higher levels of emotional distress throughout the cancer trajectory. Physicians tend to recognize and address physical symptoms from cancer and its treatment, but emotional and psychological distress is addressed less well. Furthermore, breast cancer care and treatment is typically lengthy, complex and distributed across a wide range of service providers. Younger women with breast cancer report difficulty navigating the healthcare system and feel ill informed, unprepared and dissatisfied by the lack of continuity. While there are resources that can help women be better informed and to manage symptoms, women are rarely informed of them early in the breast cancer journey, when the need is greatest.There is an urgent need to identify solutions that can be implemented at a population level and that can be accommodated within limited healthcare budgets. Education and self-management approaches that help cancer patients access appropriate knowledge and supports, and that impart skills could make a significant contribution to improving their experience and quality of life. Internet-based resources are convenient, accessible and acceptable circumventing childcare and transportation issues making it an ideal modality for YWBC who are usually more familiar with electronic communication compared to older women with breast cancer.

Active coping early in the breast cancer journey - in contrast to taking a passive stance - predicts better adjustment and quality of life years later. Access to relevant, credible and timely health information 'empowers' individuals to cope actively and better manage their own health. Over 60% of cancer patients report using the Internet for prognostic information, to identify alternative treatment options and for symptom management. Nonetheless, too much or low quality information leads to confusion and stress, and YWBC report being bombarded with information that is not relevant or timely, and lacks age-appropriate content. YWBC also report that Internet searching is exhausting and scary. Self management (SM) approaches in cancer care have the aim to empower patients by providing knowledge, and additionally, providing skills that help persons manage the physical and emotional impacts of their disease and treatment, as well as broader life challenges that living with a disease bring. SM approaches address issues such as problem solving, finding and using community resources effectively, working with the health care team, and learning how to initiate new health promotion behaviours. SM interventions have been shown to increase knowledge, reduce fatigue and distress, improve quality of life and improve lifestyle changes such as physical activity. A well-designed website with links and self-management tools could help YWBC by pointing them to the right information at the right time, by ensuring that content addresses the specific knowledge and support needs of younger women, and is based in current knowledge. We previously demonstrated that web-based professionally led support helped YWBC survivors who reported high levels of satisfaction and benefits including improved knowledge, mood, hope, and relief of burden. However, YWBC's needs were highest at the time of diagnosis, and they reported dissatisfaction with the lack of age-specific information.

We propose to develop a supported self-management website that will orient newly diagnosed YWBC to the terrain ahead, and help them cope more skilfully and proactively. We will use a time series research design to test the hypothesis that access to this website reduces distress and enhances confidence in coping with breast cancer, in three samples of newly diagnosed YWBC.

Objective 1: Develop a Supported Self-Management Website for YWBC We will develop a website that directs YWBC to the "right information at the right time" and additionally offers guidance, skills enactment and commentary that will help women be optimally active and effective. As an example, to encourage active participation in treatment decision-making which predicts later adjustment, the site will direct YWBC to the best sites for diagnostic/medical information, and to newly-developed resources including a video with peer modelling of a good doctor-patient interview, a tip sheet on effective communication with physicians, and an engaging presentation of the evidence-supported strategy of recording the consultation. We will develop engaging, age-appropriate tools include video interviews, frequently asked questions with embedded links to information and resources, and self-directed education presentations. Modules will include but not be limited to: communicating with physicians, friends and family; problem solving; assessing and managing symptoms of emotional distress and insomnia; education about the impact of hormonal changes and fertility preservation.

Objective 2: Conduct an experiment to test the clinical promise of the website The study will be conducted at 3 sites (Women's College Hospital, Princess Margaret Hospital, and Calgary Breast Health Centre), selected among the 28 sites that are participating in the CYBCC cohort study. Prior to launching the website, a baseline comparison group of 100 newly diagnosed YWBC will be recruited. They will be assessed on a number of variables, including emotional distress and self-efficacy for coping with cancer. Four months later, emotional distress and self-efficacy will be assessed again. Following completion of the website, another cohort of 100 patients will undergo the same procedure, however these participants will have the Internet website introduced to them. The two groups will then be compared to determine if access to the website reduces the traumatic stress associated with a breast cancer diagnosis and treatment, and improves coping confidence.

ELIGIBILITY:
Inclusion Criteria:

* are diagnosed with invasive or ductal carcinoma in-situ disease
* are able to read and understand English

Exclusion Criteria:

* under 18 or over 40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Traumatic stress | 4 months
  Tramatic stress will be assessed with the Impact of Event Scale (IES), measuring intrusion and avoidance symptoms related to the diagnosis of breast cancer.

SECONDARY OUTCOMES:
Cancer Behavior Inventory | 4 months
  The Cancer Behavior Inventory will assess a) beliefs about maintaining independence and a positive attitude, b) belief in ability to participate in medical care, c) skills important for coping and stress management, and d) capacity to manage emotions in difficult situations.